CLINICAL TRIAL: NCT03098264
Title: A Cohort Study on Safety and Efficacy of Simultaneous or Staged Surgery in Complicated Hepatolithiasis
Brief Title: Safety and Efficacy of Simultaneous or Staged Surgery on Complicated Hepatolithiasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Chinese PLA General Hospital (Other); Eastern Hepatobiliary Surgery Hospital (Other); First Affiliated Hospital of Zhongshan Medical University (Other); Air Force Military Medical University, China (Other); Huaxi Hospital (Other); Tongji Hospital (Other); Union hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, feng xiaobin, Doctor, Southwest Hospital, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWHB018
Record Dates: First submitted 2017-03-20; First posted 2017-03-31 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Hepatolithiasis
MeSH Terms: interventions — Overlapping Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simultaneous surgery (Experimental): to perform surgery both on biliary stone and portal hypertension
  Interventions: Procedure: Simultaneous surgery
- Staged surgery (Active Comparator): to perform surgery on biliary stone and portal hypertension by staged surgery
  Interventions: Procedure: staged surgery

INTERVENTIONS:
Procedure: Simultaneous surgery — Simultaneous surgery in complicated hepatolithiasis
  Arms: Simultaneous surgery
Procedure: staged surgery — staged surgery in complicated hepatolithiasis
  Arms: Staged surgery

SUMMARY:
For some complicated hepatolithiasis, it is difficult to decide whether to perform surgery on biliary stone and portal hypertension simultaneously or separately by staged surgery.There's a high risk of intraoperative bleeding, postoperative liver failure and variceal bleeding for these patients.How to develop a optimized algorism of simultaneous and staged surgery is highly needed.

DETAILED DESCRIPTION:
For some complicated hepatolithiasis, it is difficult to decide whether to perform surgery on biliary stone and portal hypertension simultaneously or separately by staged surgery.There's a high risk of intraoperative bleeding, postoperative liver failure and variceal bleeding for these patients.How to develop a optimized algorism of simultaneous and staged surgery is highly needed. In this protocol, we will assign the eligible cases into two group. And then perform surgery as simultaneously or separately.By long-term follow-up,to examine the safety and advantages of each procedure.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 65 years old
* Without gender restriction
* With a favorable liver function of Child-Pugh A to B
* No contraindications to surgery and anesthesia
* Diagnosed with Hepatolithiasis and portal hypertension
* Signed informed consent.

Exclusion Criteria:

* Diffused type of Hepatolithiasis
* Impairment in liver function
* Severe disorders in vital organ
* Accompanied with tumors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
residual ratio of biliary stone | 3 months
  residual ratio of biliary stone diagnosed within 3 months

SECONDARY OUTCOMES:
postoperative complications | 6 months
  postoperative complications diagnosed within 6 months
residual lesions | 6 months
  residual lesions diagnosed within 6 months
Health economics index | 3 months
  Health economics index within 3 months
mortality | 3 months
  mortality occured within 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided